CLINICAL TRIAL: NCT03544398
Title: Comparison of Exoskeleten Assisted Gait Training With End-effector Assisted Gait Training in Spinal Cord Injury
Brief Title: Comparison of an Exoskeleten With an End-effector for Assisted Gait Training in Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erenköy Physical Therapy and Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, AYLİN SARI, MD, Erenköy Physical Therapy and Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erenkoy
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exoskeleton (Active Comparator): We will use exoskeleton type robot assisted gait training for spinal cord injury rehabilitation
  Interventions: Other: robot assisted gait training
- end-effector (Active Comparator): We will use end-effector type robot assisted gait training for spinal cord injury rehabilitation
  Interventions: Other: robot assisted gait training
- conventional physiotherapy (Placebo Comparator)
  Interventions: Other: robot assisted gait training

INTERVENTIONS:
Other: robot assisted gait training — we use two types of robot assisted gait training and we will compare two groups.

SUMMARY:
Aim is to compare exoskeleton assisted gait training with end-effector assisted gait training in Spinal Cord Rehabilitation

DETAILED DESCRIPTION:
It was planned to evaluate patients aged between 18 and 80 years who will admit to the robotic rehabilitation program due to spinal cord injury. Patients will divide into three groups as Exoskeleton, End-effector and conventional therapy. Exoskeleton and End-effector group will receive robotic therapy 4 days a week besides conventional treatment for 6 weeks. All groups will be evaluated at the start and end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of spinal cord injury Applying to the hospital for a rehabilitation program

Exclusion Criteria:

Inadequate body weight (obesity) Severe contractures Bone instability ( nonstable spinal cord fracture, and severe osteoporosis) Circulation problems Cardiac nonconformity Open wounds on the lower extremities or in the body where they will come into contact with the orthosis Uncoordinated, psychotic or aggressive patients Serious cognitive disorders Long-term infusion therapy Hip, knee, ankle arthrodesis Epilepsy Disproportionate limb or vertebrae, such as bone cartilage dysplasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
FAC | Change from baseline FAC class to 6th week of therapy
  functional ambulational classification scale
6MWT | Change from baseline 6MWT class to 6th week of therapy
  6 minute walking test
10MWT | Change from baseline 10MWT class to 6th week of therapy
  10 meter walking test

SECONDARY OUTCOMES:
ASIA | Change Of ASIA scale from the beginnig to the 6th week of the therapy
  ASIA impairment scale
SCIM | Change Of SCIM from the beginnig to the 6th week of the therapy
  Spinal cord independence measure

CONTACTS AND LOCATIONS:
Overall Officials: unsal SARI, Study Chair — Dr.
Locations (1):
- Aylin Sari, Istanbul, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No